CLINICAL TRIAL: NCT01823445
Title: XyliMelts Ability to Reduce Mutans Streptococci in Adults With the Perception of Dry Mouth
Brief Title: Xylitol Disk Use in Adults With Dry Mouth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Peter Milgrom, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: XM2013
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Mutans Streptococci; Xerostomia
Keywords: Xylitol; Dental caries
MeSH Terms: conditions — Xerostomia; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xylitol disk (Experimental): Daily use of 8 disks containing 0.5 grams xylitol each for two weeks. The disks adhere to gum tissue with a food grade adhesive backing and slowly dissolve. The disks are applied one on each side of the mouth in the morning after breakfast, again at midday, and four are applied, two on each side, at bedtime.
  Interventions: Other: Xylitol disk

INTERVENTIONS:
Other: Xylitol disk
  Other Names: XyliMelts

SUMMARY:
The purpose of this study is to demonstrate whether decay causing bacteria are reduced when adhesive xylitol disks are used intraorally three times a day for two weeks in adults with dry mouth.

DETAILED DESCRIPTION:
Xylitol,an FDA approved sugar substitute, has been shown to reduce tooth decay. Patients who experience dry mouth may be more susceptible to dental decay because they lack the protection provided by an adequate flow of saliva. These patients are likely to have high levels of the decay causing bacteria, mutans streptococci.

The purpose of this research is to test the ability of a novel xylitol delivery vehicle to reduce mutans streptococci in patients with dry mouth over a two week period. The delivery vehicle is a slowly dissolving xylitol disk (lozenge) that adheres to soft tissues inside the mouth. Participants will place disks on both sides of the mouth three times a day.

ELIGIBILITY:
Inclusion Criteria:

* Adults 21 years old or older
* Daily use of at least 2 prescription medications known to cause dry mouth
* Current report of dry mouth

Exclusion Criteria:

* Antibiotic use in the last month
* Topical oral antimicrobial (e.g. Chlorhexidine rinse) use in the last month
* Change in medication or dose within the last month
* Use of mouthwash within the last week
* Use of lozenges or chewing gum with 500 mg or more of xylitol on a habitual basis
* History of gastrointestinal disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mutans streptococci levels | One week
  Change in mutans streptococci levels from Baseline to one week.
Mutans streptococci levels | Two weeks
  Change in mutans streptococci levels from Baseline to two weeks.

SECONDARY OUTCOMES:
GRIX measure of xerostomia | One week
  Change in Groningen Radiotherapy-Induced Xerostomia (GRIX) quality of life questionnaire assessing xerostomia symptoms from Baseline to one week.
GRIX measure of xerostomia | Two weeks
  Change in Groningen Radiotherapy-Induced Xerostomia (GRIX) quality of life questionnaire assessing xerostomia symptoms from Baseline to two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, School of Dentistry, Regional Clinical Dental Research Center, Seattle, Washington, United States